CLINICAL TRIAL: NCT03565289
Title: PRospective Prostate biOmarker Study (PROPOSe)
Brief Title: PRospective Prostate biOmarker Study
Acronym: PROPOSe
Status: Completed | Type: Observational
Sponsor: ProteoMediX AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PROPOSe_1
Record Dates: First submitted 2018-06-07; First posted 2018-06-21 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Indication for Prostate Biopsy Due to Suspected Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — During a routine blood draw an additional tube of blood will be taken for the study.

SUMMARY:
• Correlation of a glycoprotein panel with prostate biopsy outcome and PCa aggressiveness

DETAILED DESCRIPTION:
The main objective of this study is to correlate a glycoprotein panel with prostate biopsy outcome, i.e. distinguishing PCa from benign prostatic conditions as well as high-grade cancer. The quantities of the two protein analytes cathepsin D (CTSD) and thrombospondin 1 (THBS1) are measured in human serum samples. In combination with percent free PSA (%fPSA), the results are correlated with prostate biopsy outcome. The potential future benefit of using this glycoprotein panel is to validate positive tPSA tests in men with negative digital rectal examination (DRE) and enlarged prostates to reduce the need for undergoing a biopsy, thereby reducing unnecessary biopsies and potentially predicting high-grade disease.

ELIGIBILITY:
Inclusion Criteria:

* Male patient between 45 and 80 years old.
* tPSA between 2 and 10 ng/ml
* Prostate volume >=35 ml
* Non-suspicious DRE for prostate cancer
* Scheduled for prostate biopsy
* Patient must give written informed consent

Exclusion Criteria:

* Patient not undergoing biopsy of the prostate
* Prior prostate biopsy within the last 12 months
* Transurethral resection of the prostate (TURP) in the last 5 years
* Patients with known acute or chronic prostatitis/cystitis or other known prostate abnormalities
* Patient taking 5-alpha-reductase inhibitor
* Any other prior treatment of the prostate (cryoablation, hifu, ire, radiation therapy, alcohol instillation, etc.)

Ages: 45 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for prostate biopsy at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of PCA | 6 months
  Correlation of the glycoprotein panel algorithm with histological diagnosis of PCa
Aggressiveness of PCA | 6 months
  Correlation of the glycoprotein panel algorithm with diagnosis of significant (Gleason Score ≥7) PCa
Diagnosis of PCA | 12 months
  Correlation of the glycoprotein panel algorithm with histological diagnosis of PCa
Aggressiveness of PCA | 12 months
  Correlation of the glycoprotein panel algorithm with diagnosis of significant (Gleason Score ≥7) PCa

OTHER OUTCOMES:
Glycoprotein panel algorithm | After 12 months
  Refinement of the glycoprotein panel algorithm
Additional Biomarkers | After 12 months
  Correlation of additional biomarkers (e. g. olfactomedin 4 (OLFM4), intercellular adhesion molecule 1 (ICAM1), hypoxia up-regulated protein 1(HYOU1) and metallopeptidase inhibitor 1 (TIMP1)) with histological diagnosis of PCa

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Steuber, Prof. Dr., Principal Investigator — Martiniklinik am UKE gGmbH
Locations (11):
- Austria (2):
  - Ordensklinikum Linz, Linz, Upper Austria
  - Medizinische Universität Innsbruck, Innsbruck
- Rigshospitalet, Copenhagen, Denmark
- Germany (8):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Malteser Krankenhaus Bonn/Rhein-Sieg, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Frankfurt, Frankfurt
  - Martini Klinik am UKE GmbH, Hamburg
  - Marien-Hospital Herne, Herne
  - Daikonie Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No